CLINICAL TRIAL: NCT03179150
Title: Clinical Validation of a CAD System for the Automated Identification of Pulmonary Metastases in Oncological Patients - CADM5L
Brief Title: Clinical Validation of the M5L Lung CAD
Status: Completed | Type: Observational
Sponsor: Candiolo Cancer Institute - IRCCS (Other)
Responsible Party: Principal Investigator, Alberto Traverso, PhD, Candiolo Cancer Institute - IRCCS
Other Study IDs: 35/2017 CADM5L
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Lung Cancer Metastatic
Keywords: computer-aided diagnosis; Web; Cloud computing; lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oncological patients with extra-thoracic cancer: Patients enrolled into the study performed CT either for staging, restaging or follow-up of extrathoracic malignancies.
  Interventions: Diagnostic Test: Computed Tomography

INTERVENTIONS:
Diagnostic Test: Computed Tomography — CT scans were performed on a 128 detector rows CT scanner (Somatom Definition Flash Siemens Medical Systems, Erlangen, Germany) as in routine clinical practice in the centre

SUMMARY:
To compare the diagnostic performance and time efficiency of Computer-Aided Detection (CAD) assisted reading for the identification of pulmonary nodules in chest Computed Tomography (CT) from oncological patients with that of unassisted reading.

DETAILED DESCRIPTION:
The main aim of this study is to compare the diagnostic performance of CAD assisted interpretation with that of unassisted reading in the detection of lung metastases in consecutive patients staged for extrathoracic malignancies. This study also aims at validating a new Web/Cloud based workflow for the use of CAD systems in clinical practice, not requiring installation of additional software or hardware and potentially representing a cost-effective CAD solution for clinical facilities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed extra-thoracic neoplasm

Exclusion Criteria:

* More than 10 nodules
* Severe pulmonary fibrosis
* Diffuse bronchiectasis
* Extensive inflammatory consolidation
* Massive pleural effusion
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Between September 2015 and March 2016, 237 consecutive patients (123 men, 52%) with an average age of 62 (range 21-90 years), were enrolled in this retrospective observational single centre study. Patients enrolled into the study performed CT either for staging, restaging or follow-up of extrathoracic malignancies
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Per-patient detection sensitivity unassisted vs CAD assisted reading | 1 month after collection of data
  Comparison of the detection sensitivity between unassisted and CAD assisted reading. Per patient analysis
Per-lesion detection sensitivity unassisted vs CAD assisted reading | 1 month after collection of data
  Comparison of the detection sensitivity between unassisted and CAD assisted reading. Per-lesion analysis. Sub-analyses per nodule tissue, nodule dimension and nodule localization are included

SECONDARY OUTCOMES:
Comparison of reading time between unassisted vs CAD assisted reading | 1 month after collection of data

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Candiolo, Candiolo, Torino, Italy

IPD SHARING:
Plan to Share IPD: No